CLINICAL TRIAL: NCT05550220
Title: A Modified Cuff Leak Test and Reintubation in Mechanically Ventilated Patients: a Multicenter Randomised Controlled Trial
Brief Title: A Modified Cuff Leak Test and Reintubation in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Bing Sun, professor of treatment, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: modified CLT
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Mechanical Ventilation Complication; Weaning Failure; Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Cuff Leak Test (Experimental): The subject was placed in a semi-recumbent position.
  The subjects were placed in volume assist-control mode with the following parameters:
  * respiratory rate 15 breaths/min
  * original oxygen concentration
  * PEEP 0 cm H2O
  * the VT was set according to the subject's stable VT in the previous ventilator mode
  * inspiratory flow was set at 30 L/min with square waveform Positive cutoff value of the air leak volume was 116 mL and the air leak ratio was 0.32.
  Interventions: Diagnostic Test: Cuff Leak Test
- Usual Cuff Leak Test (Active Comparator): The subjects were placed in volume assist-control mode with the following parameters:
  * respiratory rate was adapted to patient comfort
  * original oxygen concentration and PEEP
  * the VT about 8ml/Kg IBW
  * inspiratory flow was set at 60 L/min with square waveform Positive cutoff value of the air leak volume was 110 mL and the air leak ratio was 0.15.
  Interventions: Diagnostic Test: Cuff Leak Test

INTERVENTIONS:
Diagnostic Test: Cuff Leak Test — Cuff leak test is a simple and convenient tool that can be used to predict upper-airway obstruction after extubation. The CLT is used to assess airway patency through listening for an air leak and observing changes in tidal volume (VT) after the cuff is deflated.

SUMMARY:
We hypothesized that the accuracy of the modified cuff leak test in predicting re-intubation in tracheal intubated patients is better than that of the conventional balloon leak test, thereby further reducing the re-intubation rate.

DETAILED DESCRIPTION:
The cuff leak test is an effective method for predicting the occurrence of upper airway obstruction in patients with endotracheal intubation after extubation, with high specificity and moderate sensitivity. However, there is still no clear and unified cuff leak test operation specification. A cohort study has proposed a modified method. When the patient is placed in a semi-recumbent position of 60 degrees and the ventilator is set to a low-flow square wave, it is more predictive than conventional methods. We hypothesized that the accuracy of the modified cuff leak test in predicting re-intubation in tracheal intubated patients is better than that of the conventional balloon leak test, thereby further reducing the re-intubation rate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Oral endotracheal intubation and mechanical ventilation > 36 hours
* Fulfilled the weaning criteria

Exclusion Criteria:

* The patient has a chest drainage tube and there is persistent air leak
* Abnormalities of the larynx: such as tumors or vocal cord paralysis
* The patient cannot maintain the semi-recumbent position
* Unconventional weaning, such as awake ECMO, etc
* Participated in the study during the hospitalization
* Patients or their relatives refused written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
fulfilled predefined criteria indicating the need for reintubation within 48 hours following extubation | 48 hours
  The incidence of fulfilled predefined criteria indicating the need for reintubation within 48 hours following extubation

SECONDARY OUTCOMES:
Reintubation within 48 hours after extubation | 48 hours
  The incidence of reintubation within 48 hours after extubation in the ICU.
Post-extubation stridor | 24 hours
  the occurrence of inspiratory stridor within 24 hours following tracheal extubation.
Invasive mechanical ventilation time before first extubation | 28 days
  Invasive mechanical ventilation time before first extubation
length of ICU | 90 days
  the length of patient staying in intensive care unit
length of hospital | 90 days
  the length of patient staying in hosptial
required reintubation within 48 hours following extubation | 48 hours
  The incidence of required reintubation within 48 hours after extubation in the ICU.

OTHER OUTCOMES:
mortality of 90 days | 90 days
  mortality of 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Bing Sun, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tang X, Gu YM, Shi Y, Li ZM, Cao R, Lu SG, Wu YB, Tao YF, Sun ZY, Yin YJ, Liu CY, Tang XB, Gan GF, Qin XJ, Yin D, Zhao HB, Liu CY, Zhang L, Fang P, Du LS, Li L, Tan H, Li M, Zuo YT, Sun B; Chao-Yang Mechanical Ventilation Study Collaboration Group. Modified Cuff Leak Test for Predicting the Risk of Reintubation in Patients With Invasive Mechanical Ventilation: A Multicenter, Single-Anonymized, Randomized Controlled Trial. Chest. 2025 Jul;168(1):119-130. doi: 10.1016/j.chest.2025.01.033. Epub 2025 Feb 6. PMID 39922534